CLINICAL TRIAL: NCT06223022
Title: How Are You Getting on? Nurse-led Proactive Telephone Follow-up With Patients After Completion of Primary Cancer Treatment Increases Their Sense of Security and Well-being
Brief Title: Nurse-led Proactive Telephone Follow-up With Patients After Completion of Primary Cancer Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Department of Nursing
Record Dates: First submitted 2023-12-04; First posted 2024-01-25 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Receiving regular telephone nurse-led support
  Interventions: Behavioral: Proactive nurse-led telephone follow-up
- Control (No Intervention): Receiving care as usual

INTERVENTIONS:
Behavioral: Proactive nurse-led telephone follow-up — An intervention nurse call the patients regularly with predetermined intervals and give support
  Arms: Intervention

SUMMARY:
The goal of this randomized study is to test and evaluate nurse-led telephone follow-up intervention in patients primarily curatively treated for breast cancer, colorectal cancer, and prostate cancer.

The main question aims to answer:

Does this nurse-led telephone follow-up improve patients' quality of life? Participants in both groups will be asked to fill in questionnaires regularly. The intervention group will get a telephone follow-up at predetermined intervals, while the control group will get the care as usual.The investigators will compare intervention and control groups to see if predetermined regular nurse-led telephone follow-up improves quality of life.

DETAILED DESCRIPTION:
The hypothesis is that nurse-led telephone follow-up will improve the quality of life in patients primarily curatively treated for breast cancer, colorectal cancer, and prostate cancer.

Participants in both groups will respond to a survey regularly during one year from inclusion. The intervention group will get a telephone follow-up at predetermined intervals (1, 3, 6, 9, 12 months) while the control group will get the care as usual. The usual care means that no proactive support is offered to patients from health care while they wait for follow-up, but patients are of course allowed to contact health care if they needed.

Participants in both groups are asked to respond on a survey concerning their quality of life, feelings of anxiety and depression, perception of illness, and experienced symptoms and discomfort regarding to cancer. Additionally, the number of visits at the health care during the waiting for follow-up will be collected from both group.

ELIGIBILITY:
Inclusion Criteria:

* Being primarily curatively treated for breast, colorectal-, or prostate cancer

Exclusion Criteria:

* no adjuvant treatment
* no cognitive impairment
* no known alcohol or other misuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patients' reported Quality of life | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) The questionnaire consists of 30 items. The QLQ-C30 is composed of both multi-item scales and single-items measures and includes five functional scales, three symptom scales, a global health status /QoL(quality of life) scale, and six single items.
  Twenty-eight items are answered on a four-point Likert scale with response option labeled "Nor at all", "A little", "Quite a bit" and "Very Much". The last two questions have a seven point scale, ranging from 1 ("Very Poor") to seven ("Excellent"). Higher score for a functional scale represents a high/healthy level of functioning, a high score for the global health status represents a high QoL but a high score for a symptom scale/item represents a high level of symptomatology/problems. The minimum in values is 0, and maximum in values is 100.

SECONDARY OUTCOMES:
Patients' reported anxiety and depression | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by the Hospital Anxiety and Depression Scale (HADS) and consist of 14 items designed to measure anxiety and depression in patients' in somatic care. The scale is intended to measure and/or detect changes in anxiety and depressive symptoms in patients who are not in psychiatric care. HADS consists of seven statements for each sub-scale: HADS anxiety and HADS depression, where minimum is 0-21 for each sub scale. The higher scores indicates worse outcome.
Patients' reported quality | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by EQ-5-D-5L. The EuroQol-5 dimension- 5 levels (EQ-5D-5L) descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five response levels: "no problem", "slight problems", "moderate problems", "severe problems" and "unable to/extreme problems". The last question is an EQ Visual Analogue Scale (VAS) assesses the overall current health, i.e., a quantitative measure of the patient's perception of their overall health. The lower score on the five specific dimensions indicate better outcome, while the higher score on the VAS scale indicate higher overall current health.
Patients' perceptions of illness | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by The Brief Illness Perception Questionnaire (B- IPQ). The questionnaire has a total of nine items where the first eight questions are rated on a 0-10 scale. An overall score from eight questions are summed (range 0-80) and a higher number indicates a more threatening illness perception. However each item is representing a dimension and can be used so.
Patients' experiences of breast cancer related to body image, sexual functioning, systemic therapy side effects and symptoms | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by The European Organisation for Research and Treatment of Cancer Quality of Life -The Breast Cancer module (EORTC QLQ-BR23).
  The Breast Cancer module is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-BR23 incorporates five multi-item scales to assess body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss.
  All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
Patients' experiences of colorectal cancer related to symptoms and side effects of treatment and diagnosis. | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by The European Organisation for Research and Treatment of Cancer Quality of Life - The Colorectal Cancer Module (EORTC QLQ-CR29).
  The European Organisation for Research and Treatment of Cancer Quality of Life - The Colorectal Cancer Module (EORTC QLQ-CR29) is a supplementary questionnaire module to be employed in conjunction QLQ-C30, and incorporates 4 multi-item scales and 19 single-items assessing a range of symptoms and problems common among patients with colorectal cancer.
  All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problems.
Patients' experiences of prostata cancer related to symptoms and side effects of treatment and diagnosis. | Baseline, 3 months, 6 months and 12 months from inclusion
  Measured by The European Organisation for Research and Treatment of Cancer Quality of Life -The Prostata Cancer module (EORTC QLQ-PR25). The QLQ-PR25 is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30 and incorporates five multi-item scales to assess sexual activity, sexual functioning, urinary symptoms, bowel symptoms, and hormonal treatment-related symptoms. In addition, one single item assesses incontinence aid.
  All of the scales and single-item measures range in score from 0 to 100. A high score for the Sexual Activity and Sexual Functioning scales represents a high level of functioning, whereas a high score for the Urinary, Bowel, and Hormonal Treatment-Related symptoms scales and Incontinence Aid item represents a high level of symptomatology or problems.

OTHER OUTCOMES:
Health-care consumption | Through study completion, an average of 1 year
  Data from register (Swedish Health and Welfare Board), focusing on number of registered visits in health care during the time of study.
Sick-leave | Through study completion, an average of 1 year
  Data from register (MiDAS), focusing on registered and self-reported number of days and intervals being on sick leave related to the reported diagnosis in health care during the time of study.

CONTACTS AND LOCATIONS:
Overall Officials: Senada Hajdarevic, PhD, Principal Investigator — Umeå University
Locations (1):
- Norrlands universitetssjukhus, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No